CLINICAL TRIAL: NCT02542020
Title: Prospective Evaluation of HIV Infected Patients Followed at Evandro Chagas National Institute of Infectious Disease (INI) - Oswaldo Cruz Foundation (FIOCRUZ) Using Non-invasive Methods for Estimation of Liver Fibrosis and Steatosis
Brief Title: Prospective Evaluation of HIV Patients Using Non-invasive Methods for Estimation of Liver Fibrosis and Steatosis
Acronym: Prospec-HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 32889514.4.0000.5262
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2018-02

CONDITIONS: Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome Virus; Liver Diseases; Liver Cirrhosis; Fibrosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Liver Diseases; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Human immunodeficiency virus (HIV) infection is a major global health issue with up to 40 million people infected worldwide. Due to highly active antiretroviral therapy, mortality related to acquired immunodeficiency syndrome (AIDS) has been reducing in the last decades. However, liver disease remains as an important cause of severe complications and death.

Hepatic fibrosis progression is the main responsible for liver-related outcomes in HIV-positive patients. Co-infection by hepatitis B (HBV) or hepatitis C virus (HCV) is highly prevalence in HIV patients. Chronic viral co-infection induces faster liver fibrosis progression compared to mono-infected HIV. However, published data have been reporting presence of significant liver fibrosis in HIV without HBV or HCV infection. This might be related to direct action of HIV in hepatocytes or association with others factors, such as non-alcoholic fatty liver disease (NAFLD). NAFLD is associated with metabolic factors, such as obesity and type-2 diabetes mellitus. However, antiretroviral drugs may induce abnormal body fat distribution (lipodistrophy) and insulin resistance playing an important role on this process. Liver biopsy has been historically considered as the gold standard to evaluate liver injury. However, this painful method presents several limitations. Therefore, several non-invasive methods for estimation of liver fibrosis, such as biomarkers (APRI, FIB-4, FibroTest and FibroMeter) and transient elastography by Fibroscan, have been developed as an alternative to liver biopsy. The diagnostic performance and prognostic value of biomarkers and transient elastography have been validated in patients with chronic liver diseases. However, few data are available in HIV patients, especially in those without chronic viral co-infection.

Therefore, patients, medical doctors and scientific community will be beneficiated by the future application of non-invasive methods for estimation of liver injury in clinical practice in HIV patients.

DETAILED DESCRIPTION:
In HIV-positive patients with or without chronic viral hepatitis co-infection, the primary aims of this project are: (i) to estimate the prevalence and incidence of liver injury (including progression of fibrosis, necro-inflammatory activity and steatosis) and to report the normal values of non-invasive methods in HIV population; (ii) to validate the diagnostic performance of non-invasive methods using a method without a gold standard (Latent Class Analysis); (iii) to validate the prognostic value of non-invasive markers to predict overall mortality and liver-related outcomes and (iv) to correlate liver injury with nutritional status. The secondary aim will be the constitution of a cohort of HIV patients, with or without chronic viral hepatitis co-infection for long-term follow-up of severe outcomes.

This prospective cohort study has been approved by the Local Ethical Committee (CAAE: 32889514.4.0000.5262) and it has been enrolling patients from June 2015 at the Evandro Chagas National Institute of Infectious Diseases - Oswaldo Cruz Foundation (INI - FioCruz), Rio de Janeiro, Brazil. A total of 2,000 patients will be included in this study during the next 5 years. This project aims to report the prevalence and incidence of liver disease in a representative sample of HIV patients with and without chronic viral hepatitis co-infection. In addition, the risk factors associated to presence and progression of liver fibrosis and steatosis will be identified and an innovative non-invasive management for estimation of liver injury in HIV patients will be validated.

Patients have been submitted at the same day to the following procedures: (i) clinical examination (anthropometric and demographic characteristics), (ii) blood sample collection (for blood analysis, calculation of biomarkers and stockage of samples), (iii) transient elastography (with M and XL probes by a single experienced operator (>2,000 examinations) and (iv) nutritional status (bioelectrical impedance and 24h diet recall).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Age >= 18 years

Exclusion Criteria:

* Auto-immune hepatitis
* Primary biliary cirrhosis
* Primary sclerosing cirrhosis
* Extra-hepatic cholestasis
* Acute viral hepatitis
* Hepatic ischemia
* Hepatic metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected by HIV with or without chronic viral hepatitis
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of stage of fibrosis and grade of steatosis in patients infected by HIV | change of fibrosis stage and steatosis grade from baseline at 5 years
  Staging of liver fibrosis and quantification of steatosis using non-invasive methods and correlation with risk factors

SECONDARY OUTCOMES:
Prognostic value of non-invasive methods | up to 5 years
  Evaluation of the prognostic value of non-invasive methods for prediction of severe outcomes and mortality
Prevalence of liver fibrosis | up to 3 years
  Estimation of liver fibrosis by non-invasive methods
Prevalence of liver steatosis | up to 3 years
  Estimation of liver steatosis by non-invasive methods
Diagnostic performance of non-invasive methods | up to 3 years
  Evaluation of diagnostic accuracy (sensitivity and specificity) of non-invasive methods using the Latent Class Analysis
Nutritional status | From date of inclusion until the date of first documented alteration on nutritional status, assessed up to 5 years
  Evaluation of the nutritional status by bioelectrical impedance and 24h diet recall
Progression of liver fibrosis | From date of inclusion until the date of first documented progression of liver fibrosis, assessed up to 5 years
  Estimation of liver fibrosis by non-invasive methods
Progression of liver steatosis | From date of inclusion until the date of first documented progression of liver steatosis, assessed up to 5 years
  Estimation of liver steatosis by non-invasive methods

CONTACTS AND LOCATIONS:
Overall Officials: Valdilea G Veloso, PhD, Principal Investigator — Oswaldo Cruz Foundation; Beatriz Grinsztejn, PhD, Principal Investigator — Oswaldo Cruz Foundation
Locations (1):
- Evandro Chagas National Institute of Infectious Diseases, Rio de Janeiro, Rio de Janeiro/RJ, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yanavich C, Perazzo H, Li F, Tobin N, Lee D, Zabih S, Morata M, Almeida C, Veloso VG, Grinsztejn B, Aldrovandi GM. A pilot study of microbial signatures of liver disease in those with HIV mono-infection in Rio de Janeiro, Brazil. AIDS. 2022 Jan 1;36(1):49-58. doi: 10.1097/QAD.0000000000003084. PMID 34873092
- [Derived] Yanavich C, Pacheco AG, Cardoso SW, Nunes EP, Chaves U, Freitas G, Santos R, Morata M, Veloso VG, Grinsztejn B, Perazzo H. Diagnostic value of serological biomarkers for detection of non-alcoholic fatty liver disease (NAFLD) and/or advanced liver fibrosis in people living with HIV. HIV Med. 2021 Jul;22(6):445-456. doi: 10.1111/hiv.13060. Epub 2021 Feb 2. PMID 33529485
- [Derived] Perazzo H, Cardoso SW, Yanavich C, Nunes EP, Morata M, Gorni N, da Silva PS, Cardoso C, Almeida C, Luz P, Veloso VG, Grinsztejn B. Predictive factors associated with liver fibrosis and steatosis by transient elastography in patients with HIV mono-infection under long-term combined antiretroviral therapy. J Int AIDS Soc. 2018 Nov;21(11):e25201. doi: 10.1002/jia2.25201. PMID 30394678